CLINICAL TRIAL: NCT04154228
Title: Non-invasive Evaluation of Lymphoma Patients Based on Artificial Intelligence and PET/MRI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TASMC-19-ES-0556-CTIL
Record Dates: First submitted 2019-10-29; First posted 2019-11-06 (Actual); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Lymphoma; Non Hodgkin Lymphoma; Follicular Lymphoma
Keywords: Lymphoma; Non Hodgkin Lymphoma; Follicular Lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Non-Hodgkin; Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lymphoma Patients (Experimental)
  Interventions: Diagnostic Test: PET/MR scan

INTERVENTIONS:
Diagnostic Test: PET/MR scan — Patients will undergo 18F-FDG PET/CT scans before therapy initiation, interim after 2/3 treatment cycles and end of treatment after therapy completion, as part of their routine evaluation, as well as additional follow-up scans, as clinically indicated and requested by referring physicians. Given signed written informed-consent forms, patients will undergo at each time point, immediately after completion of PET/CT, a PET/MR scan, following the same single injection of 18F-FDG. Standard preparation and acquisition protocols for FDG PET imaging will be employed.
  PET/MR imaging will include conventional sequences as T1, T2, diffusion weighted imaging, and advanced vascular imaging (DCE-MRI).

SUMMARY:
18F-FDG PET/MR imaging protocol integrating advanced MR vascular imaging sequences, along with computerized quantitative methods for data analysis, is expected to serve as an objective tool for assessment of lymphoma patients. The aim of this prospective study is to develop an automatic artificial intelligence-based tool for the assessment of early response to treatment and evaluation of residual masses in patients with lymphoma. Specific objectives are:

1. To evaluate the added value of 18F-FDG PET/MRI compared with PET/CT in imaging lymphoma.
2. To optimize PET/MR imaging protocol for lymphoma assessment.
3. To develop an automated tool for staging patients with lymphoma.
4. To develop an automated method for early prediction of response to therapy and prognosis in patients with lymphoma.
5. To develop an automated non-invasive tool for discriminating benign from active residual masses at end of treatment in patients with lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. patients with newly diagnosed hodgkin's, aggressive non-hodgkin's and follicular lymphoma (for whom the PET/CT is the imaging modality of choice)/
2. Patients aged 18 years or older of both sexes.
3. Patients treated at Tel-Aviv Sourasky Medical center.

Exclusion Criteria:

1. pregnancy,
2. contraindication to MRI or to intravenous gadolinium injection.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-12-10 (Estimated); Primary Completion 2020-01-10 (Estimated); Study Completion 2021-12-10 (Estimated)

PRIMARY OUTCOMES:
Patients that preform 18F-FDG PET/MRI and the routinely PET/CT | 1 year
  Patients that preform 18F-FDG PET/MRI and the routinely PET/CT, and the investigators optimize PET/MRI imaging protocol, and to develop an automated artificial intelligence-based tool for assessment of early response to treatment in patients with lymphoma.

IPD SHARING:
Plan to Share IPD: Undecided